CLINICAL TRIAL: NCT06928194
Title: Reliability of the Kinovea System in the Study of Spatiotemporal Gait Parameters in Multiple Sclerosis: a Pilot Study.
Brief Title: Reliability of Kinovea in Gait Assessment in Multiple Sclerosis: a Pilot Study.
Acronym: KV-MS
Status: Completed | Type: Observational
Sponsor: University of Cadiz (Other)
Collaborators: Hospital Universitario Virgen Macarena (Other)
Responsible Party: Principal Investigator, Antonio Gil Centeno, Physiotherapist, student of a master's degree in Neurological Physiotherapy, University of Cadiz
Other Study IDs: SICEIA-2025-000557
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis; Gait Disorders, Neurologic
Keywords: Multiple Sclerosis; Gait Disorders, Neurologic; Kinovea; GAITRite
MeSH Terms: conditions — Multiple Sclerosis; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The objective of this observational study is to determine whether the Kinovea video analysis tool is valid and reliable for analyzing spatiotemporal gait parameters in multiple sclerosis, comparing the data obtained from this system with those of the gold standard, the GaitRite system. The main question to be answered is:

Is the Kinovea system valid and reliable for analyzing spatiotemporal gait parameters in multiple sclerosis?

Participants walked across the GAITRite platform four times without shoes and four times with shoes, while being recorded by two cameras simultaneously: one recorded gait from the sagittal plane and the other from the frontal plane.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for evaluation by the NeuroLab-Lázaro gait laboratory (Seville).
* Patients who have signed informed consent prior to the test.
* Patients between 18 and 55 years of age, diagnosed with MS according to the 2017 McDonald criteria.
* Patients with an EDSS score of less than 6.5 points.
* Patients who are willing to participate in the study and who do not object to being recorded while performing the gait test and to the use of images for educational and research purposes.

Exclusion Criteria:

* Patients who use walking aids and/or orthoses.
* Patients with comorbidity or decompensated systemic disease within the last month.
* Patients who have any physical impediment (excessive fatigue) to performing the gait test, as documented in their medical records reviewed on the Diraya platform.
* Patients who have suffered a relapse within 30 days prior to the start of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young-to-middle-aged people with multiple sclerosis who maintain the ability to walk and who come to the laboratory for their scheduled checkups.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Step length (cm) | With the GAITRite system, measurement is instantaneous, while with the Kinovea system, measurement of all parameters took 2 hours for each patient.
  Distance between the two heel strike points during initial contact of opposing feet.
Stride length (cm) | With the GAITRite system, measurement is instantaneous, while with the Kinovea system, measurement of all parameters took 2 hours for each patient.
  Distance between the two heel strike points during initial contact of the same foot. Two step lengths add up to one stride length.
Support base (cm) | With the GAITRite system, measurement is instantaneous, while with the Kinovea system, measurement of all parameters took 2 hours for each patient.
  Distance between the midpoints of the heels of two consecutive steps
Cadence (steps/min) | With the GAITRite system, measurement is instantaneous, while with the Kinovea system, measurement of all parameters took 2 hours for each patient.
  Number of steps taken during a given period
Walking speed (cm/s) | With the GAITRite system, measurement is instantaneous, while with the Kinovea system, measurement of all parameters took 2 hours for each patient.
  Time taken to walk a known distance

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Luque Moreno, Study Director — University of Seville
Locations (1):
- NeuroLab-Lázaro, Seville, Sevilla, Spain